CLINICAL TRIAL: NCT06481748
Title: The Batman Project: Can Unpredictability Foster Prosocial Behaviour Through Increased Awareness?
Brief Title: Unleashing Unpredictability: The Batman Project and Its Impact on Prosocial Behavior and Awareness
Status: Not yet recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Pagnini, Professor, Catholic University of the Sacred Heart
Other Study IDs: 33/24
Record Dates: First submitted 2024-06-20; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Social Behavior
Keywords: mindfulness; attention; Batman; awareness; prosociality
MeSH Terms: conditions — Social Behavior | interventions — lolal protein, Drosophila

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Batman — The investigators foresee several teams engaged throughout the day to ensure greater variability, each team will consist of three students for the experimental condition (Batman; "pregnant girl", observer) and two students for the control condition ("pregnant girl" and observer), plus the presence in both cases of a member of the research team. The 'pregnant girl' will be properly prepared and equipped with a sponge prosthesis to simulate pregnancy. In addition, the subject dressed as Batman must be prepared to play the role in a natural and non-invasive manner. During this phase, the student observers collaborating in the study will carefully record the behavior of the passengers in the underground.

SUMMARY:
The proposed study is an observational investigation that aims to examine the impact of an unexpected and unusual event on prosociality within the Milan metro. The event is the simple presence, in the underground car, of a student wearing a Batman suit. The main objective is to assess whether or not the presence of the unusual event influences prosocial behaviour towards a student pretending to be pregnant. During the study, the student, equipped with a sponge prosthesis to simulate a pregnancy will board the underground. She will be asked not to interact with anyone, but to simply look at her phone. In the experimental condition, an individual dressed as Batman will enter the carriage (through a different door than the one used by the student). In the control condition, on the other hand, no one will show up in costume. In addition, the observer will try to gather information on the reason for this prosocial behaviour, noting down the answer given.

ELIGIBILITY:
Inclusion Criteria:

* Being a passenger in the metro

Exclusion Criteria:

* Metro too crowded
* Seats available

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: -All metro passengers present at the time of the experiment are potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2024-06-21 (Estimated); Primary Completion 2024-09-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Prosocial behavior | 5 minutes
  A person in the metro leave their spot to the pregnant lady

SECONDARY OUTCOMES:
Awareness | 5 minutes
  A person dressed as batman enters the metro

IPD SHARING:
Plan to Share IPD: No
No identifying data will be stored.

REFERENCES:
- [Derived] Pagnini F, Grosso F, Cavalera C, Poletti V, Minazzi GA, Missoni A, Bogani L, Bertolotti M. Unexpected events and prosocial behavior: the Batman effect. Npj Ment Health Res. 2025 Nov 3;4(1):57. doi: 10.1038/s44184-025-00171-5. PMID 41184421